CLINICAL TRIAL: NCT04233814
Title: A Randomized, Double-Blind, Placebo-Controlled, Ph 1a, First-in-Man, Single Ascending Dose & Multiple Ascending Dose Safety, Tolerability and PK Study of a Caveolin-1-Scaffolding-Protein-Derived Peptide (LTI-03) in Healthy Adult Subjects
Brief Title: Safety, Tolerability and Pharmacokinetic Study of LTI-03 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rein Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: LTI-03-1001
Record Dates: First submitted 2020-01-12; First posted 2020-01-18 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: The first part of the study will follow a Single Ascending Dose design. Subjects receive a single dose of double-blind study medication (investigational medicinal product LTI-03 or placebo) on Day 1.
  For each dose level cohort, two eligible sentinel subjects will be randomized in a 1:1 ratio to receive active:placebo study medication.
  If no tolerability issues are observed by the Investigator within 48 hours post-dose, dosing will commence for the remaining six subjects in the cohort, who will be randomized in a 5:1 ratio to receive active:placebo study medication.
  The second part of the study will follow a Multiple Ascending Dose design. Subjects receive double-blind study medication (LTI-03 or placebo) once-daily from Day 1 to Day 14.
  For each dose level cohort, eight eligible subjects will be randomized in a 6:2 ratio to receive active:placebo study medication.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The Sponsor, Investigator, and study personnel working on behalf of the Investigator and Sponsor will remain blinded.
  Study medication will be dispensed by unblinded pharmacy staff to study staff in a blinded manner. Other than the pharmacist(s), all study staff will remain blinded to study medication assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (9):
- Placebo (Sham Comparator): Matching placebo is a micronized lactose powder administered by inhalation through a dry powder inhaler (DPI)
  Interventions: Drug: Placebo
- SAD Cohort 1 (Experimental): LTI-03 20 mg delivered qd x 1 day via DPI
  Interventions: Drug: Caveolin-1-Scaffolding-Protein-Derived Peptide (LTI-03)
- SAD Cohort 2 (Experimental): LTI-03 40 mg delivered qd x 1 day via DPI
  Interventions: Drug: Caveolin-1-Scaffolding-Protein-Derived Peptide (LTI-03)
- SAD Cohort 3 (Experimental): LTI-03 80 mg delivered qd x 1 day via DPI
  Interventions: Drug: Caveolin-1-Scaffolding-Protein-Derived Peptide (LTI-03)
- MAD Cohort 1 (Experimental): LTI-03 dose at 20mg once daily x 14 days via DPI
  Interventions: Drug: Caveolin-1-Scaffolding-Protein-Derived Peptide (LTI-03)
- MAD Cohort 2 (Experimental): LTI-03 dose at 40mg once daily x 14 days via DPI
  Interventions: Drug: Caveolin-1-Scaffolding-Protein-Derived Peptide (LTI-03)
- MAD Cohort 3 (Experimental): LTI-03 dose at 2.5 mg once daily x 14 days via DPI
  Interventions: Drug: Caveolin-1-Scaffolding-Protein-Derived Peptide (LTI-03)
- MAD Cohort 4 (Experimental): LTI-03 dose at 5 mg once daily x 14 days via DPI
  Interventions: Drug: Caveolin-1-Scaffolding-Protein-Derived Peptide (LTI-03)
- MAD Cohort 5 (Experimental): LTI-03 dose at 5 mg twice daily x 14 days via DPI
  Interventions: Drug: Caveolin-1-Scaffolding-Protein-Derived Peptide (LTI-03)

INTERVENTIONS:
Drug: Caveolin-1-Scaffolding-Protein-Derived Peptide (LTI-03) — LTI-03, a Caveolin-1 scaffold protein-derived 7-amino acid peptide to be administered as a dry powder by inhalation through a dry powder inhaler.
  Arms: MAD Cohort 1; MAD Cohort 2; MAD Cohort 3; MAD Cohort 4; MAD Cohort 5; SAD Cohort 1; SAD Cohort 2; SAD Cohort 3
Drug: Placebo — Matching placebo is micronized lactose powder administered by inhalation through a dry powder inhaler.
  Arms: Placebo

SUMMARY:
The current study will investigate the initial safety, tolerability, and PK profile of inhaled LTI-03 in healthy volunteers. In order to minimize exposure, the study will first test single ascending doses (SAD) of LTI-03 followed by multiple ascending dose (MAD) cohorts.

Findings from this study will direct the clinical development of LTI-03 for the treatment of IPF

The study subject population will include normal healthy male and female volunteers between 18 and 55 years of age (inclusive).

Consistent with other trials involving inhaled medication, subjects must have normal pulmonary function at Screening and will be excluded if they have a history of active or recurring allergies, asthma, chronic obstructive pulmonary disease (COPD), chronic sinus drainage, chronic or acute cough or other respiratory condition deemed exclusionary by the Investigator. History of liver dysfunction or elevated bilirubin, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) values at Screening will also be grounds for exclusion.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoker (no use of tobacco products within 6 months prior to dosing) with a negative urine cotinine test at Screening or Day -1
2. Age of 18-55 years (inclusive)
3. Body mass index (BMI) of 18 - 30.5 kg/m2 (inclusive)
4. Body weight > 50 kg
5. Willing and able to provide written informed consent

Exclusion Criteria:

1. History of asthma
2. Presence of active or recurring allergies, asthma, chronic obstructive pulmonary disease (COPD), chronic sinus drainage, chronic or acute cough or other respiratory condition deemed exclusionary by the Investigator or designee
3. Pulmonary infiltrate or pneumonia within 6 months prior to dosing or acute infection within 14 days prior to dosing
4. History of significant allergy or anaphylaxis
5. Any clinically significant hematologic, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic or allergic disease (excluding hay fever), as determined by the Investigator or designee
6. Any current clinically relevant abnormalities identified by a detailed medical history, complete physical examination including blood pressure and heart rate measurement, and clinical laboratory tests (hematology, coagulation, urinalysis, clinical chemistries) at Screening or Day -1, as determined by the Investigator or designee
7. Any clinically significant illness and/or surgery within 28 days prior to dosing
8. Febrile illness within 7 days prior to dosing
9. Weight loss > 5 kg within 28 days prior to dosing
10. Clinically significant 12-lead electrocardiogram (ECG) abnormalities or vital sign abnormalities (systolic blood pressure < 90 mmHg or > 140 mmHg, diastolic blood pressure < 50 mmHg or > 90 mmHg, or heart rate < 45 beats per minute [bpm] or > 100 bpm) at Screening or Day -1, as determined by the Investigator or designee
11. History of, or existing severe, acute, chronic, and/or psychiatric medical condition(s), laboratory abnormality, or other medical concerns that may increase the risk associated with study participation or IMP administration which, in the judgment of the Investigator, would make the subject inappropriate for entry into the study
12. History of cancer with the exception of adequately treated basal cell or squamous cell carcinoma of the skin
13. Hemoglobin < lower limit of normal (LLN)
14. Abnormal liver function- alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 times the upper limit of the normal range (ULN)

    - total bilirubin > 1.5 times ULN
15. Abnormal renal function: estimated glomerular filtration rate (eGFR) (modification of diet and renal disease [MDRD]) < 55 mL/min/1.73 m2
16. Pulmonary function outside the normal range, including forced expiratory volume 1 (FEV1), forced vital capacity (FVC) each < 80% of predicted or FEV1/FVC ratio of ≤ 0.7 at Screening
17. Inability to use study inhaler device appropriately.
18. Positive test results for human immunodeficiency virus (HIV) HIV-1/HIV-2 antibodies, hepatitis B surface antigen (HBsAG) or hepatitis C virus antibody (HCV-AB) Concurrent Intake of Other Substances
19. History of alcohol abuse within one year prior to Screening or regular use of alcohol of ≥ 14 units of alcohol per week for females and ≥ 21 units of alcohol for males (1 unit = 150 mL wine, 360 mL beer or 45 mL of 40% alcohol) within 6 months prior to dosing or a positive urine alcohol test at Screening or Day -1
20. History of drug abuse or misuse within 5 years prior to dosing or a positive urine drug test at Screening or Day -1
21. Inability or unwillingness to abstain from alcohol or any drug of abuse for 48 hours prior to the first dose until completion of the Day 8 visit for the SAD and Day 21 visit for the MAD
22. Exposure to any live vaccines within 28 days prior to dosing
23. Treatment with an investigational product within 30 days or 5 half-lives (whichever is longer) prior to dosing
24. Use of prescription or non-prescription medications and dietary supplements within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study medication. Herbal supplements must be discontinued 28 days prior to dosing. Approved medications taken for contraception are permitted.
25. Positive serum pregnancy test in female subjects
26. Female subjects who are lactating
27. Female subjects of childbearing potential (FOCBP) and men with partners of childbearing potential who do not agree to use an acceptable form of contraception for the duration of study treatment and for at least 90 days after the last dose of study medication. Male subjects who do not agree to refrain from donating sperm during this same period.
28. Not eligible to receive study medication within 2 weeks of receiving a COVID-19 vaccination, including an initial, second, or booster injection.

NOTE: Female who is surgically sterile or post-menopausal for at least 12 months with follicle stimulating hormone (FSH) > 30 mIU/ml, are not considered to be of childbearing potential.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAE) | up to 49 days
  Incidence of TEAE by system-organ class and dose group as assessed by the Toxicity Grading Scale for Healthy Adult Volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Devinda Weeraratne, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Belfast, United Kingdom